CLINICAL TRIAL: NCT00716599
Title: Effectiveness and Safety of Training in Fever Case Management Incorporating Rapid Diagnostic Tests (RDTs) for Malaria at Peripheral Health Centers in Uganda
Brief Title: Training in Fever Case Management With Rapid Diagnostic Tests (RDTs) for Malaria in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Exxon Mobil (Industry); Makerere University (Other); Uganda Malaria Surveillance Project (Other); National Institutes of Health (NIH) (NIH); Doris Duke Charitable Foundation (Other)
Responsible Party: Heidi Hopkins, MD, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EM-036
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Malaria; Fever
Keywords: malaria; diagnosis; rapid diagnostic test; rapid diagnostic tests; fever case management; training; fever case management in malaria-endemic areas
MeSH Terms: conditions — Malaria; Fever; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Health centers continue with standard-of-care empiric case management
- RDT training (Experimental): Health centers randomly selected to receive training and RDTs, for use in routine patient case management
  Interventions: Device: training in use of rapid diagnostic tests (RDTs) for malaria

INTERVENTIONS:
Device: training in use of rapid diagnostic tests (RDTs) for malaria — training program and introduction of RDTs for use in case management of patients presenting for routine care at government health centers
  Arms: RDT training

SUMMARY:
Malaria remains one of the most devastating infectious diseases in the world. Despite the potential for serious adverse outcomes with each episode of malaria, most cases in endemic areas are diagnosed on clinical grounds alone. Even the simple technique of light microscopy, the gold standard for malaria diagnosis, is inaccessible to most individuals in resource-poor malarious areas. New diagnostic methods that are practical for limited health-care settings are urgently needed. Immunochromatographic rapid diagnostic tests (RDTs) for malaria are easy to use, require little infrastructure or expertise, show good accuracy, and are increasingly advocated for routine use in malaria-endemic areas. A major challenge now is to implement RDTs effectively in typical African clinical settings. We plan to evaluate the clinical effectiveness and safety of a training curriculum incorporating RDT use in peripheral government health centers in Uganda. Results from this study will provide evidence for scale-up of RDT implementation in Uganda, as planned by the Uganda Ministry of Health from mid-2008, as well as in other sub-Saharan African countries.

The aim of this study is to evaluate the clinical effectiveness and safety of a basic training program incorporating RDTs, as compared with standard-of-care presumptive treatment, for the management of patients who present with suspected malaria at peripheral health centers in Uganda. Our hypothesis is that training in fever case management and RDT use will allow health center staff to reduce unnecessary antimalarial prescriptions without compromising patient outcomes, compared with the current practice of presumptive antimalarial therapy for all febrile patients.

ELIGIBILITY:
Inclusion Criteria:

* all outpatients at participating health centers

Exclusion Criteria:

* patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14000 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To compare changes in the proportion of patients prescribed any antimalarial therapy between health centers with and without an RDT training intervention. | point of care

SECONDARY OUTCOMES:
To compare changes in the proportion of patients with an inadequate response to initial therapy between health centers with and without an RDT training intervention. | 5 days after initial clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Hopkins, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Uganda Malaria Surveillance Project, Kampala, Uganda

REFERENCES:
- See also: research collaboration website — http://www.muucsf.org